CLINICAL TRIAL: NCT04742517
Title: A Phase 1 Combined Single and Multiple Ascending Intravenous Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MA-0217 in Healthy Adult Subjects and Healthy Elderly Subjects
Brief Title: A Study of MA-0217 (ASP1128) in Healthy Adult Subjects and Healthy Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 1128-CL-0101
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteers
Keywords: MA-0217; Healthy Volunteers; Pharmacokinetics; ASP1128
MeSH Terms: interventions — ASP1128

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Single ascending dose of ASP1128 (Experimental): Participants (6 for each cohort) will receive a single dose of ASP1128.
  Interventions: Drug: ASP1128
- Single ascending dose of Placebo (Placebo Comparator): Participants (2 for each cohort) will receive a single dose of matching Placebo.
  Interventions: Drug: Placebo
- Multiple ascending dose of ASP1128 (Experimental): Participants (9 for each cohort) will receive daily doses of ASP1128 for 7 consecutive days.
  Interventions: Drug: ASP1128
- Multiple ascending dose of Placebo (Placebo Comparator): Participants (3 for each cohort) will receive matching Placebo for 7 consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP1128 — Intravenous
  Other Names: MA-0217
  Arms: Multiple ascending dose of ASP1128; Single ascending dose of ASP1128
Drug: Placebo — Intravenous
  Arms: Multiple ascending dose of Placebo; Single ascending dose of Placebo

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability of single ascending intravenous doses of ASP1128 in healthy adult male and female subjects and multiple ascending intravenous doses of ASP1128 in healthy adult male and female subjects and healthy elderly male and female subjects.

This study will also evaluate the pharmacokinetics and the effect on the QT interval using Fridericia's correction formula (QTcF) in these subjects.

DETAILED DESCRIPTION:
After a screening period of up to 28 days prior to study drug administration, eligible participants will be residential for a single period of 5 days/4 nights in Part 1: single ascending dose, and 11 days/10 nights in Part 2 multiple ascending dose.

Part 1 is composed of 6 parallel cohorts (cohorts 1.1 to 1.6) and up to 2 optional cohorts (cohorts 1.7 and 1.8) of 8 healthy adult male and female subjects in each cohort. If the data from cohorts 1.1 to 1.6 are not sufficient to characterize safety, tolerability and pharmacokinetics, up to 2 optional cohorts (cohorts 1.7 and 1.8) may be added.

Part 2 is composed of 4 parallel cohorts (cohorts 2.1 to 2.4) and 1 optional cohort (cohort 2.5) of 12 healthy adult male and female subjects in each cohort and 1 cohort (cohort 2.6) of 12 healthy elderly male and female subjects. Dosing of the elderly cohort (cohort 2.6) will commence after having established the safety and tolerability of the corresponding dose tested in cohorts 2.1 to 2.5. If the data from cohorts 2.1 to 2.4 are not sufficient to characterize safety, tolerability and pharmacokinetics, 1 optional cohort (cohort 2.5) may be added.

ELIGIBILITY:
Inclusion Criteria:

* For adult subjects (cohorts 1.1 to 1.8 and cohorts 2.1 to 2.5):

  * Subject is a healthy adult male or female subject 18 to 55 years of age, inclusive at screening.
  * Subject has a body mass index (BMI) range of 18.5 to 32.0 kg/m^2, inclusive and weighs at least 50 kg at screening.
* For elderly subjects (cohort 2.6):

  * Subject is a healthy elderly male or female subject ≥ 65 years of age at screening.
  * Subject has a BMI range of 18.5 to 32.0 kg/m^2, inclusive and weighs at least 50 kg at screening.
* Subject is considered an adult according to local regulation at the time of signing informed consent.
* Female subject must either be of nonchildbearing potential:

  * Postmenopausal (defined as at least 1 year without any menses for which there is no other obvious pathological or physiological cause) prior to screening, or
  * Documented surgically sterile (e.g., hysterectomy, bilateral salpingectomy or bilateral oophorectomy), OR, if of childbearing potential:
  * Agree not to try to become pregnant during the study and for 28 days after the final study drug administration
  * Have a negative blood pregnancy test at screening and a negative urine pregnancy test on day -1
  * If heterosexually active, agree to consistently use 1 form of highly effective birth control starting at screening and throughout the study period and for 28 days after the final study drug administration
* Female subject must agree not to breastfeed starting at screening and throughout the study period and for 28 days after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period and for 28 days after the final study drug administration.
* A sexually active male subject with female partner(s) who is(are) of childbearing potential is eligible for the study if:

  * Agree to use a male condom starting at screening and continue throughout study treatment and for 28 days after the final study drug administration.
  * If the male subject has not had a vasectomy or is not sterile, their female partner(s) is(are) utilizing 1 form of highly effective birth control starting at screening and continue throughout study treatment and for 28 days after the male subject receives their final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the study period and for 28 days after the final study drug administration.
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner(s) is(are) breastfeeding throughout the study period and for 28 days after the final study drug administration.
* Subject agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Subject has received investigational drug within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Subject has any condition which makes the subject unsuitable for study participation.
* Female subject who has been pregnant within 6 months prior to screening or breastfeeding within 3 months prior to screening.
* Subject has a known or suspected hypersensitivity to ASP1128 or any components of the formulation used.
* Subject has had previous exposure with ASP1128.
* Subject has unsuitable or difficult venous access to support the intravenous infusion(s) and/or required blood draws.
* Subject has any of the liver function tests (LFTs; aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase [ALP], gamma-glutamyl transferase and total bilirubin [TBL]) above the upper limit of normal (ULN) at screening or on day -1. In such a case, the assessment may be repeated once.
* Subject has total creatine kinase (CK) > 1.5 × ULN or cardiac troponin I above the ULN at day -1.
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema, or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies) prior to study drug administration.
* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (noncutaneous) infection within 1 week prior to day -1.
* Subject has any clinically significant abnormality following the physical examination, electrocardiogram (ECG) and protocol-defined clinical laboratory tests at screening or on day -1.
* Subject has a mean pulse < 45 or > 90 bpm; mean systolic blood pressure (SBP) > 140 mmHg; mean diastolic blood pressure (DBP) > 90 mmHg (measurements taken in triplicate after subject has been resting in the supine position for at least 5 minutes; pulse will be measured automatically) at screening or on day -1. For elderly subjects the following criteria apply: SBP > 160 mmHg, DBP > 100 mmHg. If the mean blood pressure exceeds the limits above, 1 additional triplicate can be taken.
* Subject has a mean QT interval using Fridericia's correction formula (QTcF) interval of > 430 msec (for males) and > 450 msec (for females) at screening or on day -1. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG can be taken.
* Subject has used any prescribed or nonprescribed drugs (including vitamins, natural and herbal remedies, e.g., St. John's Wort) in the 2 weeks prior to study drug administration, except for occasional use of acetaminophen (up to 2 g/day), hormonal contraceptives and hormone replacement therapy.
* Subject has used any peroxisome proliferator-activated receptor (PPAR) ligands such as fibrates and thiazolidinediones, including self-medication obtained via the internet, in the 4 weeks prior to study drug administration.
* Subject has smoked or has used tobacco-containing products and nicotine or nicotine-containing products in the past 6 months prior to screening.
* Subject has a history of consuming > 14 units of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/substance abuse within past 2 years prior to screening (Note: 1 unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits/hard liquor) or the subject tests positive for alcohol or drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and opiates) at screening or on day -1.
* Subject has used any drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and opiates) within 3 months prior to day -1.
* Subject has used any inducer of metabolism (e.g., barbiturates and rifampin) in the 3 months prior to day -1.
* Subject has had significant blood loss, donated ≥ 1 unit (450 mL) of blood or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to day -1.
* Subject has a positive serology test for hepatitis B surface antigen (HBsAg), hepatitis B core (HBc) antibodies, hepatitis A virus (HAV) antibodies (immunoglobulin M [IgM]), hepatitis C virus (HCV) antibodies or antibodies to human immunodeficiency virus (HIV) type 1 and/or type 2 at screening.
* Subject is an employee of Astellas, Mitobridge or designated contract research organization (CRO).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-09-07 (Actual); Study Completion 2018-09-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) in Part 1 | Up to Day 16
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.
  In order to identify any events that may be associated with study procedures and could lead to a change in the conduct of the study, AEs will be collected even if the subject has not received study drug treatment.
Number of participants with laboratory value abnormalities and/or AEs in Part 1 | Up to Day 16
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and/or AEs in Part 1 | Up to Day 16
  Number of participants with potentially clinically significant vital sign values.
Number of participants with electrocardiogram (ECG) abnormalities and/or AEs in Part 1 | Up to Day 16
  Number of participants with potentially clinically significant 12-ECG values.
Number of participants with real-time cardiac monitoring (cardiac telemetry) abnormalities and/or AEs in Part 1 | On Day 1
  Number of participants with potentially clinically significant cardiac telemetry values.
Number of participants with AEs in Part 2 | Up to Day 19
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.
  In order to identify any events that may be associated with study procedures and could lead to a change in the conduct of the study, AEs will be collected even if the subject has not received study drug treatment.
Number of participants with laboratory value abnormalities and/or AEs in Part 2 | Up to Day 19
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and /or AEs in Part 2 | Up to Day 19
  Number of participants with potentially clinically significant vital sign values.
Number of participants with ECG abnormalities and/or AEs in Part 2 | Up to Day 19
  Number of participants with potentially clinically significant 12-ECG values.

SECONDARY OUTCOMES:
Part 1: Pharmacokinetics (PK) of ASP1128 in plasma: Area under the concentration-time curve (AUC) from the time of dosing extrapolated to time infinity (AUCinf) | Up to 72 hours post-dose on Day 1
  AUCinf will be recorded from the PK plasma samples collected.
Part 1: PK of ASP1128 in plasma: AUC from the time of dosing to the last measurable concentration (AUClast) | Up to 72 hours post-dose on Day 1
  AUClast will be recorded from the PK plasma samples collected.
Part 1: PK of ASP1128 in plasma: percentage of AUCinf due to extrapolation from time of the last measurable concentration to time infinity (AUCinf(%extrap)) | Up to 72 hours post-dose on Day 1
  AUCinf(%extrap) will be recorded from the PK plasma samples collected.
Part 1: PK of ASP1128 in plasma: maximum concentration (Cmax) | Up to 72 hours post-dose on Day 1
  Cmax will be recorded from the PK plasma samples collected.
Part 1: PK of ASP1128 in plasma: total systemic clearance after intravenous dosing (CL) | Up to 72 hours post-dose on Day 1
  CL will be recorded from the PK plasma samples collected.
Part 1: PK of ASP1128 in plasma: time of maximum concentration (tmax) | Up to 72 hours post-dose on Day 1
  Tmax will be recorded from the PK plasma samples collected.
Part 1: PK of ASP1128 in plasma: terminal elimination half-life (t1/2) | Up to 72 hours post-dose on Day 1
  T1/2 will be recorded from the PK plasma samples collected.
Part 1: PK of ASP1128 in plasma: volume of distribution during terminal elimination phase after intravenous dosing (Vz) | Up to 72 hours post-dose on Day 1
  Vz will be recorded from the PK plasma samples collected.
Part 1: PK of ASP1128 in plasma: volume of distribution at steady state determined after intravenous dosing (Vss) | Up to 72 hours post-dose on Day 1
  Vss will be recorded from the PK plasma samples collected.
Part 1: PK of ASP1128 in urine: cumulative amount of study drug excreted into urine from time of dosing up to the collection time of the last measurable concentration (Aelast) | Up to 72 hours post-dose on Day 1
  Aelast will be recorded from the PK urine samples collected.
Part 1: PK of ASP1128 in urine: percentage of study drug dose excreted into urine from time of dosing up to the collection time of the last measurable concentration (Aelast%) | Up to 72 hours post-dose on Day 1
  Aelast(%) will be recorded from the PK urine samples collected.
Part 1: PK of ASP1128 in urine: cumulative amount of study drug excreted into urine from time of dosing extrapolated to time infinity (Aeinf) | Up to 72 hours post-dose on Day 1
  Aeinf will be recorded from the PK urine samples collected.
Part 1: PK of ASP1128 in urine: percentage of study drug dose excreted into urine from time of dosing extrapolated to time infinity (Aeinf(%)) | Up to 72 hours post-dose on Day 1
  Aeinf(%) will be recorded from the PK urine samples collected.
Part 1: PK of ASP1128 in urine: renal clearance (CLR) | Up to 72 hours post-dose on Day 1
  CLR will be recorded from the PK urine samples collected.
Part 2 (first dose): PK of ASP1128 in plasma: AUC from the time of dosing to 24 hours (AUC24) | Up to 24 hours post-dose on Day 1
  AUC24 will be recorded from the PK plasma samples collected. This will be replaced with ACU12 in case of twice daily dosing.
Part 2 (first dose and last dose): PK of ASP1128 in plasma: Cmax | Up to 24 hours post-dose on Day 1 and up to 72 hours post-dose on Day 7
  Cmax will be recorded from the PK plasma samples collected.
Part 2 (first dose and last dose): PK of ASP1128 in plasma: tmax | Up to 24 hours post-dose on Day 1 and up to 72 hours post-dose on Day 7
  Tmax will be recorded from the PK plasma samples collected.
Part 2 (last dose): PK of ASP1128 in plasma: area under the concentration time curve from the time of dosing to the start of the next dosing interval (AUCtau) | Up to 24 hours post-dose on Day 7
  AUCtau will be recorded from the PK plasma samples collected
Part 2 (first dose): PK of ASP1128 in plasma: AUCinf | Up to 24 hours post-dose on Day 1
  AUCinf will be recorded from the PK plasma samples collected.
Part 2 (first and last dose): PK of ASP1128 in plasma: CL | Up to 24 hours post-dose on Day 1 and up to 72 hours post-dose on Day 7
  CL will be recorded from the PK plasma samples collected.
Part 2 (last dose): PK of ASP1128 in plasma: peak trough ratio (PTR) | Up to 72 hours post-dose on Day 7
  PTR will be recorded from the PK plasma samples collected.
Part 2 (last dose): PK of ASP1128 in plasma: accumulation ratio calculated using AUC (Rac(AUC)) | Up to 24 hours post-dose on Day 1 and up to 24 hours post-dose on Day 7
  Rac(AUC) will be recorded from the PK plasma samples collected
Part 2 (first and last dose): PK of ASP1128 in plasma: t1/2 | Up to 24 hours post-dose on Day 1 and up to 72 hours post-dose on Day 7
  T1/2 will be recorded from the PK plasma samples collected.
Part 2 (first and last dose): PK of ASP1128 in plasma: Vz | Up to 24 hours post-dose on Day 1 and up to 72 hours post-dose on Day 7
  Vz will be recorded from the PK plasma samples collected.
Part 2 (first and last dose): PK of ASP1128 in plasma: Vss | Up to 24 hours post-dose on Day 1 and up to 72 hours post-dose on Day 7
  Vss will be recorded from the PK plasma samples collected.
Part 2 (last dose): PK of ASP1128 in urine: cumulative amount of study drug excreted into urine from the time of dosing to the start of the next dosing interval (Aetau) | Up to 24 hours post-dose on Day 7
  Aetau will be recorded from the PK urine samples collected.
Part 2 (last dose): PK of ASP1128 in urine: percentage of study drug dose excreted into urine from the time of dosing to the start of the next dosing interval (Aetau%) | Up to 24 hours post-dose on Day 7
  Aetau% will be recorded from the PK urine samples collected.
Part 2 (last dose): PK of ASP1128 in urine: CLR | Up to 24 hours post-dose on Day 7
  CLR will be recorded from the PK urine samples collected.
Part 2 (Dose on days 2, 4 and 6): PK of ASP1128 in plasma: concentration immediately prior to dosing at multiple dosing (Ctrough) | Pre-dose on Day 2, 4 and 6
  Ctrough will be recorded from the PK plasma samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Europe BV (APEB)
Locations (1):
- Parexel Early Phase Clinical Unit - Los Angeles, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Taniuchi Y, van Till JWO, Wojtkowski T, Toyoshima J, Koibuchi A, Sargent B, Han D. Single- and Multiple-dose Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ASP1128, a Novel Peroxisome Proliferator-activated Receptor delta Modulator, in Healthy Participants. Clin Pharmacol Drug Dev. 2023 Aug;12(8):810-818. doi: 10.1002/cpdd.1236. Epub 2023 Mar 21. PMID 36942507